CLINICAL TRIAL: NCT02531412
Title: Spironolactone Administration to Prevent Ischemic Kidney Injury in Critically Ill Cancer Patients
Acronym: SPIROCAN
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Dr. Bertha Cordova-Sanchez, MD, Instituto Nacional de Cancerologia de Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CEI/993
Record Dates: First submitted 2015-08-19; First posted 2015-08-24 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Critically Ill; Cancer
Keywords: Acute kidney injury; Critically ill cancer patients; Spironolactone
MeSH Terms: conditions — Critical Illness; Neoplasms; Acute Kidney Injury | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spironolactone (Experimental): Spironolactone 25 mg PO daily for three days. During five days investigators will collect values of plasma creatinine, sodium, potassium, blood ureic nitrogen, vital signs and urinary output.
  Interventions: Drug: Spironolactone
- Placebo (Placebo Comparator): Placebo 25mg PO daily for three days During five days investigators will collect values of plasma creatinine, sodium, potassium, blood ureic nitrogen, vital signs and urinary output.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone — After a major surgery event a time 0, 24h and 48h
  Other Names: Aldactone
  Arms: Spironolactone
Drug: Placebo — After a major surgery event a time 0, 24h and 48h
  Arms: Placebo

SUMMARY:
Acute kidney injury frequently affects cancer patients. The main cause of acute kidney injury is ischemic damage caused by transient decrease in renal blood flow, followed by blood flow restoration and accompanying reperfusion injury (ischemia-reperfusion injury. Several studies, mainly in animal models have tried to establish spironolactone role on kidney injury induced by ischemia-reperfusion injury. It has been demonstrated in renal transplant recipients that the administration of spironolactone can prevent oxidative stress and is safe. The group of cancer patients with states capable of producing tissue hypoperfusion (hypovolemic shock, heart failure, major surgery, use of anesthetics) are at increased risk of developing acute renal ischemia-reperfusion injury.

The investigators hypothesis is that spironolactone may be useful in preventing acute renal injury when administered during the first six hour of renal ischemia-reperfusion insult.

The purpose of this study is to determine the utility of spironolactone administered after an ischemic renal insult (major surgery) to prevent acute kidney injury in critically cancer patients.

Investigators propose a pilot study, randomized, double blind, placebo controlled trial, approved by the local ethical committee, to compare the efficacy of spironolactone to prevent acute kidney injury in patients after major surgery. Investigators will include 12 patients in spironolactone group (25mg daily for three days) and 12 patients in placebo group.

DETAILED DESCRIPTION:
Acute kidney injury frequently affects cancer patients, with an estimated annual risk of 17.5% after cancer diagnosis. In critically ill cancer patients, acute kidney injury incidence varies between 12 to 49%, and between 9 and 32% need renal replacement therapy. In this last group of patients, acute kidney injury frequently occurs as part of multiple organic failure and is associated with a mortality rate of 53 to 93%, as well as an increment in costs and days of hospitalization.

The main cause of acute kidney injury is ischemic damage caused by transient decrease in renal blood flow, followed by blood flow restoration and accompanying reperfusion injury (ischemia-reperfusion injury.

The decrease on renal blood flow is followed by an increment of aldosterone, this hormone acts on epithelial cells through mineralocorticoid receptors in several tissues, including heart and kidneys. In kidneys, aldosterone promotes sodium absorption and potassium excretion.

The decrease in renal blood flow is a strong stimulus for aldosterone secretion. This hormone has non-genomic actions on smooth muscle cells and vascular endothelium, causing vasoconstriction, interleukin and oxygen reactive species generation, and beta-transforming growth factor (TGF BETA) mediated fibrosis, among others.

At renal level, it has been demonstrated that mineralocorticoid receptor blockade can prevent proteinuria and glomerulosclerosis development in animal models of chronic kidney disease. Moreover, in chronic kidney disease patients with proteinuria, spironolactone addition to angiotensin converting enzyme inhibitors (ACEI), reduces proteinuria in 42% without a higher risk of hyperkalemia.

Several studies, mainly in animal models have tried to establish spironolactone role on kidney injury induced by ischemia-reperfusion injury.

In an acute and chronic cyclosporine (CyA) nephrotoxicity rat model, spironolactone administration prevented kidney injury associated to afferent arteriole vasoconstriction.

In an animal ischemia-reperfusion model produced by renal artery clipping, spironolactone administration one (Sp1), two (Sp2) or three (Sp3) days before ischemic insult resulted in better renal plasmatic flow and creatinine clearance, and prevented histopathological ischemic lesions. Spironolactone administration stimulated nitric oxide production and prevented lipid peroxidation and caspase 3 mediated apoptotic injury.

To determine aldosterone blockade effects after ischemic injury, a new group of animals received spironolactone at 0, 3, 6 and 9 hours after IR insult. Spironolactone administration up to 6 hours after IR insult prevented histologic kidney tubular damage. KIM-1 mRNA levels did not augmented in 0 and 3 hour groups, suggesting that spironolactone administration up to three hours after renal ischemic injury prevented kidney damage.

Considering that IR injury is the principal etiologic agent on acute kidney injury in renal transplant patients, in 2013, a pilot double blinded clinical trial included 20 living kidney transplants divided in spironolactone (25mg per day) or placebo groups, receiving the drug one day before and three days after renal transplant surgery. It was observed that in spironolactone prophylactically treated patients, urinary levels of hydrogen peroxide were inferior at the fifth day compared to placebo group, however, there were no differences in serum creatinine levels nor in other urinary biomarkers (KIM-1, IL-18, HSP-72). In this trial, no patient developed potassium levels higher than 6mEq/dL and there was only one patient in each group with serum potassium higher than 5mEq/L, demonstrating that spironolactone administration was safe.

The group of cancer patients with states capable of producing tissue hypoperfusion (hypovolemic shock, heart failure, major surgery, use of anesthetics) are at increased risk of developing acute renal ischemia-reperfusion injury.

The investigators hypothesis is that spironolactone may be useful in preventing acute renal injury when administered during the first six hour of renal ischemia-reperfusion insult.

The purpose of this study is to determine the utility of spironolactone administered after an ischemic renal insult (major surgery) to prevent acute kidney injury in critically cancer patients.

Investigators propose a pilot study, randomized, double blind, placebo controlled trial, approved by the local ethical committee, to compare the efficacy of spironolactone to prevent acute kidney injury in patients after major surgery. Investigators will include 12 patients in spironolactone group (25mg daily for three days) and 12 patients in placebo group. During five days investigators will collect values of plasma creatinine, sodium, potassium, blood ureic nitrogen, vital signs and urinary output.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU in the immediate postoperative period (first 24 hours) of major surgery, defined as involving general anesthesia, ventilation, opening of large cavities (cranial, thoracic, abdominal).
* Patients with informed consent signed by them or their responsible relative.
* Patients who are likely to survive at least 48 hours after admission to the ICU.
* Patients who have measured "baseline" creatinine before UCI admission, in the last three months.

Exclusion Criteria:

* Patients who have contraindications for enteral medications.
* Patients who have acute kidney injury at the time of admission.
* Patients on renal replacement therapy prior to ICU admission.
* Patients with previous diagnosis of chronic kidney disease G3b stage.
* Patients with plasma potassium greater than 5.1mEq/L.
* Hypersensitivity to spironolactone.
* Septic shock.
* Obstructive uropathy.
* Renal transplantation.
* Postoperative period of nephrectomy.
* Pregnancy.
* Known adrenal insufficiency.
* Patients requiring a higher dose of norepinephrine 0.1mcg/kg/min for more than an hour to maintain mean arterial pressure equal to or greater than 70mmHg even after receiving fluid resuscitation.
* Patients requiring the administration of inhibitors of angiotensin-converting enzyme (ACE) for its management.
* Patients requiring an increase of 25% or more of the dose of norepinephrine to maintain mean arterial pressure equal of greater than 70mmHg during follow up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Acute kidney injury by 0.3 creatinine elevation | 48 hours
  Elevation of creatinine to 0.3mg/dL above baseline in the last 48 hours
Acute kidney injury by 1.5 times creatinine elevation | 48 hours
  Elevation of baseline creatinine 1.5 times above baseline
Acute kidney injury by urinary output | 48 hours
  Decreased urine output less than 0.5ml/kg/hr over a period of 6 continuous hours somewhere during the first 48 hours monitoring, after admission to the intensive care unit

SECONDARY OUTCOMES:
Hyperkalemia | Up to 5 days
  Serum potassium above 5.1mE/L

CONTACTS AND LOCATIONS:
Overall Officials: Bertha M Cordova-Sanchez, MD, Principal Investigator — Instituto Nacional de Cancerologia, Columbia
Locations (1):
- Nacional Cancer Institute, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No